CLINICAL TRIAL: NCT02826733
Title: Evaluation of the Implementation of the Hemispheric Dominance During Development : Electrometabolic and Hemodynamics Study in the Newborn Born Premature or Term
Brief Title: Evaluation of the Implementation of the Hemispheric Dominance During Development
Acronym: HEMISPHERENOR
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Centre Hospitalier Universitaire, Amiens (Other)
Responsible Party: Sponsor
Other Study IDs: PI08-DR-WALLOIS
Record Dates: First submitted 2016-07-05; First posted 2016-07-11 (Estimated); Last update posted 2023-02-08 (Actual); Status verified 2023-02

CONDITIONS: Neuroimaging
Keywords: preterm infants; term infants; hemispheric dominance
MeSH Terms: interventions — Electroencephalography; Magnetic Resonance Imaging

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective

GROUPS / COHORTS (2):
- Normal: Every child meet the age criteria and without ductus arteriosus persistence ultrasound or detectable neurological disorders after clinical, neurophysiological and radiological (ETF , Scanner, MRI).
  EEG NIRS MRI
  Interventions: Device: Electroencephalogram (EEG); Device: Near Infra Red Spectroscopy (NIRS); Device: magnetic resonance imaging (MRI)
- cerebral neurological disease: Group of children meeting the criteria of age and having a detectable neurological disease after clinical, neurophysiological and radiological (ETF , Scanner, MRI) The children present either convulsions or a cerebrovascular accident or a neurological pain . Each condition being verified by a pathological electroencephalogram .
  EEG NIRS MRI
  Interventions: Device: Electroencephalogram (EEG); Device: Near Infra Red Spectroscopy (NIRS); Device: magnetic resonance imaging (MRI)

INTERVENTIONS:
Device: Electroencephalogram (EEG)
Device: Near Infra Red Spectroscopy (NIRS)
Device: magnetic resonance imaging (MRI)

SUMMARY:
Many cognitive functions in human are based on asymmetric brain networks. For most adults, language is processed largely by the left hemisphere while other auditory treatments, such as voice recognition are rather based on the right hemisphere. Many studies helped to highlight the presence of anatomical and functional asymmetries both in the first months of life. What are the causes of these imbalances? How do they develop? Are they necessary for operation or for effective learning?

The investigators would like in this work, in collaboration with applied mathematics team of Compiègne and INSERM team, to determine from which period the development of hemispheric dominance is set up for recognition of language and in which brain structure it occurs in preterm infants whose sound environment is usually very different from that of the fetus. The impact of this environment on brain development of infants and their early learning will be assessed.

ELIGIBILITY:
Inclusion Criteria:

* preterm gestational age over 26 weeks of gestation + 6 days and less than 42 weeks.
* normal group of children : A child meets the age criteria and without ductus arteriosus persistence ultrasound or detectable neurological disorders after clinical, neurophysiological and radiological (ETF , Scanner, MRI).
* Group of children meet the age criteria and with cerebral neurological pathology detectable after clinical, neurophysiological and radiological (ETF , Scanner, MRI).

Exclusion Criteria:

* severe congenital malformation
* Any refusal of a parent .
* Children with severe impairment of the general condition and vital functions
* Children with dermatitis of the face or scalp
* Children treated with ventilation High Frequency (HFO )
* Presence of intravenous access on the scalp ( preventing the realization of the ETF , EEG or NIRS .

Ages: 0 Days to 10 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: The inclusion of patients in the study will be conducted in the intensive care unit and neonatal intensive care CHU Amiens .
Sampling Method: Non-Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2009-11-04 (Actual); Primary Completion 2021-11-03 (Actual); Study Completion 2024-11-03 (Estimated)

PRIMARY OUTCOMES:
discrimination of language - EEG | Day 0
  Determine at what developmental age the newborn and premature are able to discriminate language based on the results of evoked potentials obtained from the EEG signals
discrimination of language - NIRS | Day 0
  Determine at what developmental age the newborn and premature are able to discriminate language based on the results of evoked potentials obtained from the NIRS signals

CONTACTS AND LOCATIONS:
Overall Officials: Fabrice WALLOIS, MD, PhD, Principal Investigator — CHU Amiens
Locations (1):
- CHU Amiens, Amiens, France